CLINICAL TRIAL: NCT05605873
Title: Clinical, Histological and Prognostic Forms of Adenocarcinoma of the Anus
Acronym: ProCHADA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ProCHADA
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Anal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adenocarcinoma of the anus is rare. It concerns less than 10% of anal cancers and its incidence is less than 0.2/100 000 inhabitants. Its management is not consensual and is most often derived by analogy with that of adenocarcinoma of the lower rectum. This is due to the rarity but also to the diversity of anatomical (anal margin, anal canal, lower rectum), etiological (primary glandular tumors or secondary to anal fistula, primary distant tumor and/or Crohn's disease) and histological forms (mucinous, intestinal, glandular adenocarcinomas and primary or secondary Paget's disease). Most of the literature consists of small case series and simple clinical cases in which the prognosis of these subforms has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* French-speaking patient
* Patient with a diagnosis of adenocarcinoma of the anus between 01/01/2006 and 30/06/2022 in participating centers

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of adenocarcinoma of the anus between 01/01/2006 and 30/06/2022 in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of mortality at 1 year, estimated using a survival curve | Year1
  This outcome corresponds to the 1 year mortality rates after diagnosis of adenocarcinoma of the anus.
Risk of mortality at 5 years, estimated using a survival curve | Year5
  This outcome corresponds to the 5 year mortality rates after diagnosis of adenocarcinoma of the anus.

SECONDARY OUTCOMES:
Describe the various anatomical, etiological and histological forms | Year5
  This outcome corresponds to the classification of anatomical (anal margin, anal canal, lower rectum), etiological (primary glandular tumors or secondary to anal fistula, primary distant tumor and/or Crohn's disease) and histological (mucinous, intestinal, glandular adenocarcinoma and primary or secondary Paget's disease) forms.
Adaptaion of the therapeutic management according to the clinical and histological form | Year5
  This outcome corresponds to the Proposed treatments (local excision, abdominoperineal amputation, neoadjuvant treatment, adjuvant treatment, etc.) according to the clinical and histological form.
Describe their therapeutic management | Year5
  This outcome corresponds to the Proposed treatments (local excision, abdominal-perineal amputation, neoadjuvant treatment, adjuvant treatment, etc.).
Compare prognosis by clinical and histological form | Year5
  This outcome corresponds to the Mortality rate by clinical and histological form.
Search for prognostic factors of severity in all forms | Year5
  This outcome corresponds to the Prognostic factors of severity for all forms.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De PARADES, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre hospitalo-universitaire de Cochin-Port Royal, Paris

REFERENCES:
- [Background] Anwar S, Welbourn H, Hill J, Sebag-Montefiore D. Adenocarcinoma of the anal canal - a systematic review. Colorectal Dis. 2013 Dec;15(12):1481-8. doi: 10.1111/codi.12325. PMID 23809885
- [Background] Lukovic J, Kim JJ, Liu ZA, Cummings BJ, Brierley JD, Wong RKS, Ringash JG, Dawson LA, Barry A, Krzyzanowska MK, Chen EX, Hedley DW, Quereshy FA, Swallow CJ, Gryfe RN, Kennedy ED, Easson AM, Hosni A. Anal Adenocarcinoma: A Rare Entity in Need of Multidisciplinary Management. Dis Colon Rectum. 2022 Feb 1;65(2):189-197. doi: 10.1097/DCR.0000000000002281. PMID 34990422
- [Background] Wang Q, Fu J, Chen X, Cai C, Ruan H, Du J. What factors are associated with the poor prognosis of anal adenocarcinoma compared with low-lying rectal adenocarcinoma based on a population analysis: A propensity score matching study. PLoS One. 2019 Jul 30;14(7):e0219937. doi: 10.1371/journal.pone.0219937. eCollection 2019. PMID 31361759
- [Background] Yasuhara M, Beppu N, Uchino M, Ikeuchi H, Matsuda I, Hirota S, Ikeda M, Tomita N. Adverse Oncologic Outcomes of Adenocarcinoma of the Anal Canal in Patients With Crohn's Disease. Dis Colon Rectum. 2021 Apr 1;64(4):409-419. doi: 10.1097/DCR.0000000000001874. PMID 33394780
- [Background] Lee GC, Kunitake H, Stafford C, Bordeianou LG, Francone TD, Ricciardi R. High Risk of Proximal and Local Neoplasms in 2206 Patients With Anogenital Extramammary Paget's Disease. Dis Colon Rectum. 2019 Nov;62(11):1283-1293. doi: 10.1097/DCR.0000000000001487. PMID 31567917